CLINICAL TRIAL: NCT01027936
Title: An Age-Stratified Data Collection Study in Adult Males and Females, Ages 18 and Above to Establish a Normative Database Using the 3D Optical Coherence Tomography 3D OCT-1000 Mark II
Brief Title: An Age-Stratified Data Collection Study to Establish a Normative Database Using the 3D Optical Coherence Tomography 3D OCT-1000 Mark II
Status: Withdrawn | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: NDB-001
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Healthy Volunteers

SUMMARY:
To collect three dimensional retinal measurements of the optic disc and the macula lutea on healthy normal subjects using the 3D OCT-1000 Mark II for the purpose of developing a normative database that is stratified by age.

ELIGIBILITY:
Inclusion Criteria:

* Male and Females at least 18 years of age;
* Must be a member of one of the 3 ethnic groups: Caucasian, Hispanic or African American. Asians, Eastern Indians, and Native Americans have been excluded from this study;
* Signed, written informed consent obtained for the study;
* BSCVA of 20/40 or better in both eyes;
* Intraocular pressure (IOP) ≤ 21 mm Hg in both eyes.

Exclusion Criteria:

* Ocular disease;
* Cataract on slit lamp exam with a corresponding loss of BSCVA worse than 20/25;
* Corneal surface disruption precluding imaging;
* Prior ocular surgery except uncomplicated phacoemulsification or strabismus surgery;
* Prior corneal refractive surgery of any type;
* Family history of glaucoma among first generation relatives;
* Current history of an acute or chronic disease or illness that would confound the normative outcome(s) of the study;
* Current use of systemic medications that may confound the outcome of the study;
* Nystagmus or any other condition that would prevent a steady gaze during study tests or measurements;
* Current history of inflammation or infection of the eye or eyelids; injury to the eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 180 male and female volunteers from 6 centers with normal, healthy eyes form six age groups, aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2009-04-30 (Actual); Study Completion 2009-04-30 (Actual)

PRIMARY OUTCOMES:
A normative dataset containing a statistical description of expected norms of retinal nerve fiber layer (RNFL) and macula lutea thickness, stratified by age. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weinreb, M.D., Study Director — University of California, San Diego; Shiley Eye Center
Locations (6):
- United States (6):
  - Shiley Eye Center UCSD, La Jolla, California
  - Durrie Vision, Overland Park, Kansas
  - Glaucoma Associates of New York, New York, New York
  - Vitreous-Retina-Macula Consultants of New York, P.C., New York, New York
  - SUNY, New York, New York
  - Eye Institute/Medical College of WI, Milwaukee, Wisconsin